CLINICAL TRIAL: NCT02620514
Title: Assessment of Health Literacy, Medication Adherence, and a Pilot Multi-component Intervention to Improve Medication Adherence in Patients With Inflammatory Bowel Disease
Brief Title: Medication Adherence in Patients With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Heba Iskandar, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00075262
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Digestive Disease and Disorders; Inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Digestive System Diseases; Disease; Inflammation | interventions — Educational Status; Financial Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Health-literacy Assessment (No Intervention): Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants with low adherence will continue to one or more intervention groups that address needs based on the results of the survey.
- Health-literacy Assessment + Education and Reminders (Experimental): Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants with then complete a 24-week intervention aimed to improve education about inflammatory bowel disease and scheduled nurse phone call reminders.
  Interventions: Behavioral: Education and Reminders
- Health-literacy Assessment + Educational Visit (Experimental): Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will then receive education about IBD.
  Interventions: Behavioral: Educational Visit
- Health-literacy Assessment + Medication Educational Visit (Experimental): Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will then receive education regarding their medications.
  Interventions: Behavioral: Medication Educational Visit
- Health-literacy Assessment + Financial Support (Experimental): Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will then receive financial support for medications.
  Interventions: Behavioral: Financial Support

INTERVENTIONS:
Behavioral: Education and Reminders — Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will be provided education materials, and will receive scheduled educational reminder phone calls and text messages at 2,6,12, and 24 weeks from the baseline assessment.
  Arms: Health-literacy Assessment + Education and Reminders
Behavioral: Educational Visit — Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence.Participants will undergo one scheduled visit with a nurse practitioner or physician for education about inflammatory bowel disease (IBD) after the baseline assessment.
  Arms: Health-literacy Assessment + Educational Visit
Behavioral: Medication Educational Visit — Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will undergo one scheduled visit with a nurse practitioner or physician to discuss medication side effects and medication inadequacy after the baseline assessment.
  Arms: Health-literacy Assessment + Medication Educational Visit
Behavioral: Financial Support — Participants with inflammatory bowel disease (IBD) will complete health-literacy surveys to assess medication adherence. Participants will receive information about patient assistance programs, copay cards, and a scheduled meeting with a social worker or financial advisor.
  Arms: Health-literacy Assessment + Financial Support

SUMMARY:
The purpose of this is to formally assess health literacy and medication adherence in participants with Inflammatory bowel disease (IBD). The study also aims to improve medication adherence, health-related quality of life, and disease activity through a 24-week intervention.

DETAILED DESCRIPTION:
The purpose of this study is to formally assess health literacy and medication adherence in participants with Inflammatory bowel disease (IBD). The study also aims to improve medication adherence, health-related quality of life, and disease activity through a 24-week intervention that will include telephone reminders, educational materials, visits to the physician, and financial counseling.

ELIGIBILITY:
Inclusion Criteria:

* New or existing diagnosis of inflammatory bowel disease (IBD) proven via endoscopy, pathology, and radiology findings
* Maintained or started on a medication for inflammatory bowel disease at the time of enrollment
* Ability to speak English
* Good hearing
* Phone availability

Exclusion Criteria:

* Pregnancy or plans to be pregnant
* Inability to make own health care decisions
* Inability to participate in the study phone calls
* Uncontrolled psychiatric illness
* Enrollment in another clinical trial outside of the standard clinic IBD registry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Medication Possession Ratio (MPR) | 12 Weeks, End of Study (Up to 24 weeks)
  The Medication possession Rate (MPR) will be calculated as the amount of medication consumed divided by days in the interval and adherence will be defined as greater than 80%.
Change in Modified Morisky Adherence Scale-8 (MMAS-8) Score | 12 Weeks, End of Study (Up to 24 weeks)
  MMAS-8 is an 8-item scale that has been validated to measure adherence in IBD patients (scoring details are claimed as proprietary information by the scale's copyright holder).

SECONDARY OUTCOMES:
Change in Harvey Bradshaw Index (HBI) Score | 12 Weeks, End of Study (Up to 24 weeks)
  The HBI is a self-administered questionnaire that assesses IBD severity. A score of less than 5 is generally considered to represent clinical remission. A score of 8 to 9 or higher are considered severe disease.
Change in Simple Colitis Activity Index (SCAI) Score | 12 Weeks, End of Study (Up to 24 weeks)
  The SCAI is a way of scoring disease activity in Ulcerative Colitis based on six simple questions about symptoms that gives a number between 0-19 that corresponds to the severity of disease activity. This index gives more detailed information on how active disease is using a number.
Change in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score | 12 Weeks, End of Study (Up to 24 weeks)
  The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a health-related quality of life tool measuring physical, social, and emotional status. Scores range from 10-70. A lower score indicates poor quality of life while a higher score indicates greater quality of life.
Change in Hospital Anxiety and Depression Scale (HADS) Score | 12 Weeks, End of Study (Up to 24 weeks)
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale that asks participants to describe how they feel. Scores range between 0 and 21. A score of 0 to 7 is normal. A score of 8 to 10 indicates borderline depression/anxiety. A score of 11-21 indicates a case of depression/anxiety.
Change in Disease Activity Assessed by the Number of Admissions | 12 Weeks, End of Study (Up to 24 weeks)
  Individual participant data will be collected regarding the number of admissions to monitor IBD remission or progression.
Change in Disease Activity Assessed by the Number of Clinic Visits | 12 Weeks, End of Study (Up to 24 weeks)
  Individual participant data will be collected regarding the number of clinic visits to monitor IBD remission or progression.
Change in Disease Activity Assessed by the Number of Emergency Visits | 12 Weeks, End of Study (Up to 24 weeks)
  Individual participant data will be collected regarding the number of emergency room visits to monitor IBD remission or progression.
Change in Disease Activity Assessed by the Number of Surgeries | 12 Weeks, End of Study (Up to 24 weeks)
  Individual participant data will be collected regarding the number of surgeries to monitor IBD remission or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Iskandar, MD, Principal Investigator — Emory University
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States